CLINICAL TRIAL: NCT06800287
Title: Prospective Observational Study On Pharmacological Voluntary Termination Of Pregnancy: Predictors Of Pelvic Pain During Treatment
Brief Title: Pharmacological Voluntary Termination of Pregnancy: Predictors of Pelvic Pain During Treatment
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IVG - OS
Record Dates: First submitted 2024-11-28; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy Related
Keywords: pelvic pain; ivg; predictive factors; pregnancy; voluntary interruption of pregnancy; pharmacological treatment
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pharmacological treatment for voluntary termination of pregnancy is a safe and effective practice, but has as its limitation a greater need for analgesic coverage than surgical treatment. Despite this, to date there are no specific guidelines on the management of pain therapy during pharmacological voluntary termination of pregnancy and in particular on its correlation with gestational age at the time of treatment. The aim of the study is to investigate the correlation between the pain symptoms reported by the patients and the gestational age at the time of the pharmacological voluntary interruption of pregnancy and to identify the presence of possible predictive factors, in order to be able to outline the correct therapeutic management.

DETAILED DESCRIPTION:
According to the Law 194 of 1978, in Italy the voluntary interruption of pregnancy (IVG) can be requested by the woman within the first 90 days of gestation for health reasons, economic, social or family. Voluntary termination of pregnancy may be achieved by surgical or pharmacological treatment.

The surgical treatment involves hysteroaspiration associated with instrumental revision of uterine cavity (RCU).

The drug treatment involves administration of mifepristone (known as RU486), followed by approximately 48 hours after administration of prostaglandins. The World Health Organization in a 2003 publication, updated in 2012, has indicated mifepristone as one of the pharmacological treatments for IVG in the first 9 weeks of gestation. Since July 2009, the AIFA has authorised its marketing in Italy. The choice between the two treatments depends on the gestational age and the patient's preferences, after careful counselling with the gynecologist, about the risks and benefits of both procedures.

In particular, until a few months ago, pharmacological treatment was reserved in Italy exclusively for patients who required IVG within the 49° day of amenorrhea. Beyond this threshold, and within the 90 days of gestation, IVG was allowed only with surgical treatment.

The Ministry of Health on 12 August 2020 issued the circular "Guidelines on voluntary termination of pregnancy with mifepristone and prostaglandins", updating the previous one dated 24 June 2010.

Based on this update, voluntary termination of pregnancy with a pharmacological method is possible up to 63 days, equal to 9 weeks completed, gestational age.

Pharmacological treatment is allowed in adequately equipped public outpatient facilities, functionally connected to the hospital and authorised by the Region, as well as in day hospitals (DH).

Drug treatment is a safe and effective practice, but it has as its limit a greater need for analgesic coverage than surgical treatment.

Many women report it as an extremely painful experience. Despite this, there are no specific guidelines on the management of pain relief therapy in the course of pharmacological IVG and in particular on its correlation with the gestational age at the time of IVG.

The aim of this study is to investigate the correlation between the painful symptoms reported by patients and the gestational age at the time of IVG and to identify the presence of any predictive factors, in order to outline the correct therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* IVG certificate issued by the doctor and signed by the woman
* Informed consent for drug treatment
* Informed consent for the study in question
* Pregnancy in utero with ultrasound date less than or equal to 63 days

Exclusion Criteria:

* Suspected extrauterine pregnancy or adnexal masses of undefined diagnosis
* IUD in place
* Severe anaemia
* Hereditary porphyria
* Coagulopathy or ongoing treatment with anticoagulants
* Ongoing treatment with corticosteroids or adrenal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requesting a pharmacological voluntary termination of pregnancy, according to Law 194 of 1978
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Pain symptoms of patients undergoing pharmacological IVG | 48 hours after the administration of mifepristone and after an observation period of not less than 3 hours
  Assessing the pain symptoms of patients undergoing pharmacological IVG recorded according to the Visual Analog Scale (VAS) scale and the need for additional analgesic therapy (rescue dose), in relation to certain variables such as the patient's age, gestational age, anxiety trait and pre-procedure anxiety state of the patients assessed by means of scientifically validated questionnaires.
  - VAS questionnaire: 0-100 numeric scale to record the patient's pain symptoms. 0 is considered the absence of pain, ≤ 40 tolerable pain (not requiring supplementary therapy), > 40 ≤ 70 intense pain (responsive to required supplementary therapy), > 70 intolerable pain not responsive to required supplementary therapy, 100 maximum pain perceived in the patient's life.

SECONDARY OUTCOMES:
Patient satisfaction | 48 hours after the administration of mifepristone and after an observation period of not less than 3 hours
  Assessing patient satisfaction by administering a questionnaire: 0-4 numerical scale to record the patient's degree of satisfaction. It is considered 0 not at all satisfied, 1 slightly satisfied, 2 fairly satisfied, 3 very satisfied, 4 completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Seracchioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - Azienda USL di Bologna, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna